CLINICAL TRIAL: NCT04361526
Title: Pilot Study on Cytokine Filtration in COVID-19 ARDS (CytokCOVID19)
Brief Title: Pilot Study on Cytokine Filtration in COVID-19 ARDS
Acronym: CytokCOVID19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Manuel Castellà (Other)
Responsible Party: Sponsor-Investigator, Manuel Castellà, MD PhDHead of the Cardiovascular Surgery Department, Associate Professor, Principal Investigator, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCB/2020/0464
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Coronavirus Infection; Acute Respiratory Distress Syndrome; COVID
Keywords: COVID; ARDS; Coronavirus
MeSH Terms: conditions — Coronavirus Infections; Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: This is a two-branch randomized, controlled, uni-center study. Eligible patients will be randomly assigned in a 1:1 ratio to receive cytokine filtration plus standard intensive care, or standard intensive care alone
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): standard intensive care alone
- Cytokine Adsorption (Experimental): cytokine adsorption plus standard intensive care
  Interventions: Device: Cytokine Adsorption

INTERVENTIONS:
Device: Cytokine Adsorption — Cytokine adsorption will be performed through a venous hemodialysis catheter, preferably jugular or femoral. The filtration system will be established with a cytokine adsorption cartridge in an hemoperfusion system using a blood flow rate of 150 - 200 ml/min. Adsorbent therapy will last 72 hours, changing cartridges every 24 hours. Prior to start, heparinization will be stablished by a 1mg/Kg iv Na heparin bolus plus iv perfusion. Activated Partial Thromboplastin Time (aPTT) control will be performed every 6 hours, with a goal range between 60 and 80 seconds.
  Arms: Cytokine Adsorption

SUMMARY:
Background: There are no proven therapies for COVID-19 infection. COVID-19 infects the respiratory epithelium of the lower airways, causing widespread damage via cytopathic effects, resulting in severe inflammation and Pneumonitis. High local and circulating levels of cytokines, or cytokine storm, can lead to capillary leak syndrome, progressive lung injury, respiratory failure and acute respiratory distress syndrome (ARDS).

Methods: This is a pilot randomized, controlled, uni-center study testing safety and efficacy of cytokine filtration on patients with severe ARDS. Eligible patients will be randomized to 72 hours filtration or no filtration on top of the standard treatment for ARDS. Indications for randomization are patients with moderate or severe ARDS with need of ventilation support (either invasive or non-invasive), with inflammatory markers. The primary outcome will be days on mechanical ventilation (MV) support. Secondary outcomes are 30-day mortality, ICU days, need for extracorporeal membrane oxygenation (ECMO) support, duration of renal replacement therapy (RRT) and catecholamine therapies, hospital length of stay, multi-organ failure. All analysis will be done according to the intention to treat principle.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Positive revere transcription polymerase chain reaction (RT-PCR) for COVID-19 in a respiratory track sample
3. Acute (less than 36 hours) onset of moderate to severe ARDS, as defined by Berlin criteria:

   * Having pneumonia or worsening respiratory symptoms
   * Bilateral pulmonary infiltrates on chest imaging (X-ray of CT scan)
   * Pulmonary wedge pressure <18 mmHg or no clinical signs of left heart failure
   * Hypoxemia: arterial oxygen pressure/Fraction of inspired oxygen (PaO2/FiO2 ratio) <200mmHg, moderate dyspnea with signs of important respiratory workload, tachypnoea >30bpm
4. Rise of inflammatory biomarkers: C-reactive protein (CRP) >10 mg/L

Exclusion Criteria:

1. Patients with a known contraindication for anticoagulation
2. Pregnancy or breast feeding
3. Patient already included in another research study
4. Decision by a physician that involvement in the study is not in the patient's best interest
5. Failure to have patient's authorization. In case of a mechanical intubated patient, lack of authorization from a first line family member
6. Multi-organ failure
7. Patients treated with Tocilizumab at the time of start filtration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Mechanical ventilation-free days | up to 28days
  Number of ventilator-free days (VFDs) at day 28 (defined as days being alive and free from mechanical ventilation at day 28 after enrollment. For patients ventilated 28 days or longer and for ventilated subjects who die, VFD is 0

SECONDARY OUTCOMES:
30-day mortality | up to 30 days
length of ICU stay (days) | up to 30 days
length of hospital stay | up to 30 days
Duration of renal replacement and cathecolamines therapies | up to 30 days
Need for extracorporeal membrane oxygenation (ECMO) support | up to 30 days
multi-organ failure measured by the Sequential Organ Failure Assessment (SOFA) score | up to 30 days (measured on days 0, 1, 2, 3, 4, 5, 6, and the last day of mechanical ventilation)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Castellà, MD PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Naicker S, Yang CW, Hwang SJ, Liu BC, Chen JH, Jha V. The Novel Coronavirus 2019 epidemic and kidneys. Kidney Int. 2020 May;97(5):824-828. doi: 10.1016/j.kint.2020.03.001. Epub 2020 Mar 7. No abstract available. PMID 32204907
- [Background] multicenter collaboration group of Department of Science and Technology of Guangdong Province and Health Commission of Guangdong Province for chloroquine in the treatment of novel coronavirus pneumonia. [Expert consensus on chloroquine phosphate for the treatment of novel coronavirus pneumonia]. Zhonghua Jie He He Hu Xi Za Zhi. 2020 Mar 12;43(3):185-188. doi: 10.3760/cma.j.issn.1001-0939.2020.03.009. Chinese. PMID 32164085
- [Background] Sheahan TP, Sims AC, Leist SR, Schafer A, Won J, Brown AJ, Montgomery SA, Hogg A, Babusis D, Clarke MO, Spahn JE, Bauer L, Sellers S, Porter D, Feng JY, Cihlar T, Jordan R, Denison MR, Baric RS. Comparative therapeutic efficacy of remdesivir and combination lopinavir, ritonavir, and interferon beta against MERS-CoV. Nat Commun. 2020 Jan 10;11(1):222. doi: 10.1038/s41467-019-13940-6. PMID 31924756
- [Background] de Wit E, Feldmann F, Cronin J, Jordan R, Okumura A, Thomas T, Scott D, Cihlar T, Feldmann H. Prophylactic and therapeutic remdesivir (GS-5734) treatment in the rhesus macaque model of MERS-CoV infection. Proc Natl Acad Sci U S A. 2020 Mar 24;117(12):6771-6776. doi: 10.1073/pnas.1922083117. Epub 2020 Feb 13. PMID 32054787
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578